CLINICAL TRIAL: NCT03642925
Title: Efficacy of Balanced Nutrition Meal Replacement Along With a Caloric Restriction on Body Weight Control
Acronym: nutrition
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chung Shan Medical University (Other)
Responsible Party: Principal Investigator, Chin Kun Wang, Professor, Chung Shan Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CS15124
Record Dates: First submitted 2018-08-10; First posted 2018-08-22 (Actual); Last update posted 2018-08-22 (Actual); Status verified 2018-08

CONDITIONS: Obesity; Diet Modification; Nutrient; Excess
Keywords: Meal replacement; calorie restriction; body weight
MeSH Terms: conditions — Obesity; Body Weight

STUDY DESIGN:
Intervention Model Description: To evaluate the impact of a nutritionally balanced conventional meal replacement diet (rich in soy/pea protein and soluble fibers) with caloric restriction in Taiwanese obese subjects.
Masking Description: it's a Open-label clinical trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Meal replacement diet (Experimental): Obese subjects (BMI>27; n=50, male 23, female 27) were requested to replace (intervention) two meals/day (breakfast and lunch or dinner) by balanced nutritional meal replacement diet (equal to 240 kcal) for 8 weeks
  Interventions: Dietary Supplement: Meal replacement diet

INTERVENTIONS:
Dietary Supplement: Meal replacement diet — Obese subjects were requested to replace two meals/day (breakfast and lunch or dinner) by balanced nutritional meal replacement diet (equal to 240 kcal) for 8 weeks with one regular meal and make sure the daily target calorie limit should be less than 1500 kcal/day for men and 1200 kcal/day for women.

SUMMARY:
The present study was designed to evaluate the impact of a nutritionally balanced conventional meal replacement diet with caloric restriction (intervention for 8 weeks) in Taiwanese obese subjects. Various parameters like anthropometric (body weight, body fat, waist circumference), lipid profile (TC, LDL-c and TG), cardiovascular risk factors, glycemic and oxidative markers as well as renal and hepatic markers were evaluated.

DETAILED DESCRIPTION:
The present study was designed to evaluate the impact of a nutritionally balanced conventional meal replacement diet (rich in soy/pea protein and soluble fibers) with caloric restriction in Taiwanese obese subjects. Obese subjects (BMI>27; n=50, male 23, female 27) were recruited and requested to replace two meals/day (breakfast and lunch or dinner) by balanced nutritional meal replacement diet (equal to 240 kcal) for 8 weeks with one regular meal and make sure the daily target calorie limit should be less than 1500 kcal/day for men and 1200 kcal/day for women.

ELIGIBILITY:
Inclusion Criteria:

* Healthy obese subject (BMI >27)
* Aged between 20 to 80 of both genders with a desire to lose weight.

Exclusion Criteria:

* Subjects with cancer
* Hyperglycemic (diabetic)
* Hypertension,
* Stroke
* Renal dysfunction
* Cardiac or hepatic dysfunctio
* allergic to the dairy product and eating disorders
* Pregnancy, nursing (lactating), chain smokers and heavy alcoholic subjects

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2015-11-21 (Actual); Primary Completion 2016-01-21 (Actual); Study Completion 2016-03-01 (Actual)

PRIMARY OUTCOMES:
Calorie intake in obese subjects | 8 weeks
  Intervention with calorie restricted meal replacement diet for 8 weeks to check the changes in calories (Kcal)
Anthropometric parameter | 8 weeks
  Intervention with calorie restricted meal replacement diet for 8 weeks to check the change in body weight (kg)
Anthropometric parameter | 8 Weeks
  Intervention with calorie restricted meal replacement diet for 8 weeks to check the change in BMI (Kg/m2)
Cardiovascular (CV) risk factors | 8 Weeks
  Intervention with calorie restricted meal replacement diet for 8 weeks to check the changes in CV risk factor like Homocysteine (umol/L)
Glycemic markers | 8 Weeks
  Intervention with calorie restricted meal replacement diet for 8 weeks to check the changes in Glycemic marker like FBG (mg/dL)
Lipid profile | 8 weeks
  Intervention with calorie restricted meal replacement diet for 8 weeks to check the changes in total cholesterol (mg/dl)

CONTACTS AND LOCATIONS:
Locations (1):
- Chung Shan Medical University, Taichung, Taichung, Taiwan

IPD SHARING:
Plan to Share IPD: No